CLINICAL TRIAL: NCT01608204
Title: Busulfan Pharmacokinetic Analysis and GST Pharmacogenetic Profile in Adults Undergoing Hematological Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, N_Krivoy, Director Clinical Pharmacology Unit, Rambam Health Care Campus
Other Study IDs: BU/MEAdultPK/PGx1
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2012-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Pharmacokinetics; Busulfan; Polymorphism; GST; MDR-1(p-Glycoprotein); Acute Myeloid Leukemia adult patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood was used for DNA extraction
Oversight: Data Monitoring Committee: No

SUMMARY:
The correlation between Busulfan Pharmacokinetics in AML transplanted patients and their GST (A1,T1,M1 and P1), MDR-1 genetic profile. If a pre-genetic testing of those genes can be utilized as biomarkers of SOS and/or HGVHD. This study is not an interventional study it is only checking the GST gene and MDR-1 gene

DETAILED DESCRIPTION:
BU levels are largely unpredictable, patients are often exposed to the toxic effects of inappropriate drug regimens before dose modifications can be made. Although the importance of TDM cannot be over emphasized, it entails trial and error and does not allow for pre- treatment dose optimization. This study, which provides an integration of genetic and pharmacokinetic data analysis of patients preconditioned for HSCT with high dose oral BU, aims to define biomarkers predictive of poor BU metabolism and clearance to prevent potential drug toxicity.This study is not an interventional study, only investigates the GST and MDR-1 genes in correlation with the "routine" Busulfan AUC done during the preparative regimen in HSCT for AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myeloid Leukemia who are clinically selected for HSCT according to known protocols.

Exclusion Criteria:

* Unable to give informed consent

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering from AML who were selected to be treated by Hematological Stem Cell Transplantation
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
If GST and ABCB1 genes modify busulfan pharmacokinetics in AML patients who will be transplanted | end of BMT transplantation
  If individuals diagnosed with AML carrying the GSTP1 variant allele rs1695 (heterozygotes) are at risk of developing supra-therapeutic BU AUC due to lower BU clearance, and if combined polymorphisms in GSTM1 and ABCB1 (3435 or 2677) are associated with BU clearance rates and AUC.